CLINICAL TRIAL: NCT04575844
Title: Effects of Exercise and GLP-1 Agonism on Muscle Microvascular Perfusion and Insulin Action in Adults With Metabolic Syndrome
Acronym: ZQL008
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Zhenqi Liu, Professor, Division of Endocrinology and Metabolism, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 200065; R01DK125330 (NIH)
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Liraglutide; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Exercise Alone (Experimental): 24 weeks of treatment
  Interventions: Other: Exercise training
- Liraglutide Alone (Experimental): 24 weeks of treatment
  Interventions: Drug: Liraglutide
- Exercise + Liraglutide (Experimental): 24 weeks f treatment
  Interventions: Drug: Liraglutide + Exercise training

INTERVENTIONS:
Drug: Liraglutide — 24 weeks of Liraglutide
  Arms: Liraglutide Alone
Other: Exercise training — 24 weeks of Exercise training
  Arms: Exercise Alone
Drug: Liraglutide + Exercise training — 24 weeks of Liraglutide + Exercise training
  Arms: Exercise + Liraglutide

SUMMARY:
The primary objective of this study is to examine whether exercise training alone, liraglutide treatment alone or exercise training plus liraglutide treatment increases cardiac and skeletal muscle microvascular blood volume, improves vascular function of the conduit vessels, and enhances insulin's metabolic action in humans with Metabolic Syndrome. Subjects will be randomized to one of the 4 groups: control, exercise training, liraglutide treatment, and exercise + liraglutide. They will be studied at the baseline and then after 24 weeks of intervention.

DETAILED DESCRIPTION:
Our hypothesis is that sustained activation of the GLP-1 receptor with Liraglutide and exercise training each will enhance microvascular insulin responses and angiogenesis in both cardiac and skeletal muscle to increase muscle insulin delivery and action and the combination of both is more effective than either alone in adults with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥21 and ≤60 years old.
* Body mass index >25 and ≤35 kg/m2 and is weight stable (<5 kg weight change in the past 6 months). BMI is limited to ≤35 kg/m2 for easier vascular access and cardiac imaging.
* Meet 3 of 5 National Cholesterol Education Program Adult Treatment Panel III Metabolic Syndrome criteria:

  * Increased waist circumference (≥102 cm in men; ≥88 cm in women)
  * Elevated triglycerides (≥150 mg/dl)
  * Reduced HDL-cholesterol (<40mg/dl in men, <50 mg/dl in women)
  * High blood pressure (≥130 mmHg systolic or ≥85mmHg diastolic)
  * Elevated fasting glucose (≥100 mg/dl)
  * Subject may participate if on the following drugs, provided the drug doses have been stable for at least 3 months.
  * Ace inhibitor
  * ARB
  * HMG CoA reductase inhibitor
  * Beta blocker
  * Calcium channel blockers
  * Alpha-adrenergic antagonist
  * Statin

Exclusion Criteria:

* A diagnosis of any type of diabetes or history of diabetes medication use
* Recently active (>20 min of moderate/high intensity exercise, 2 times/week)
* Subjects who are smokers or who have quit smoking <5 years
* Subjects with hypertriglyceridemia (>400 mg/dl) or hypercholesterolemia (>260 mg/dl)
* Subjects with BP>160/90
* Subjects with a history of significant metabolic, cardiac, cerebrovascular, hematological, pulmonary, gastrointestinal, liver, renal, or endocrine disease or malignancy
* Pregnant (as evidenced by positive pregnancy test) or nursing women
* Subjects with contraindications to participation in an exercise training program
* Allergic to perflutren
* A prior use of Liraglutide

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular Blood Volume - change from baseline | 24 weeks
  measured at baseline and 24 weeks

SECONDARY OUTCOMES:
Augmentation Index - change from baseline | 24 weeks
  measured at baseline and 24 weeks
Flow Mediated Dilation | 24 weeks
  measured at baseline and 24 weeks
Pulse Wave Velocity | 24 weeks
  measured at baseline and 24 weeks
Post Ischemic Flow Velocity - change from baseline | 24weeks
  measured at baseline and 24 weeks
Insulin Sensitivity - change from baseline | 24 weeks
  measured at baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhenqi Liu, MD, Principal Investigator — Division of Endocrinology and Metabolism, University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] le Roux CW, Astrup A, Fujioka K, Greenway F, Lau DCW, Van Gaal L, Ortiz RV, Wilding JPH, Skjoth TV, Manning LS, Pi-Sunyer X; SCALE Obesity Prediabetes NN8022-1839 Study Group. 3 years of liraglutide versus placebo for type 2 diabetes risk reduction and weight management in individuals with prediabetes: a randomised, double-blind trial. Lancet. 2017 Apr 8;389(10077):1399-1409. doi: 10.1016/S0140-6736(17)30069-7. Epub 2017 Feb 23. PMID 28237263
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Barrett EJ, Wang H, Upchurch CT, Liu Z. Insulin regulates its own delivery to skeletal muscle by feed-forward actions on the vasculature. Am J Physiol Endocrinol Metab. 2011 Aug;301(2):E252-63. doi: 10.1152/ajpendo.00186.2011. Epub 2011 May 24. PMID 21610226
- [Background] Vincent MA, Clerk LH, Lindner JR, Klibanov AL, Clark MG, Rattigan S, Barrett EJ. Microvascular recruitment is an early insulin effect that regulates skeletal muscle glucose uptake in vivo. Diabetes. 2004 Jun;53(6):1418-23. doi: 10.2337/diabetes.53.6.1418. PMID 15161743
- [Background] Eggleston EM, Jahn LA, Barrett EJ. Hyperinsulinemia rapidly increases human muscle microvascular perfusion but fails to increase muscle insulin clearance: evidence that a saturable process mediates muscle insulin uptake. Diabetes. 2007 Dec;56(12):2958-63. doi: 10.2337/db07-0670. Epub 2007 Aug 24. PMID 17720897
- [Background] Chai W, Wang W, Liu J, Barrett EJ, Carey RM, Cao W, Liu Z. Angiotensin II type 1 and type 2 receptors regulate basal skeletal muscle microvascular volume and glucose use. Hypertension. 2010 Feb;55(2):523-30. doi: 10.1161/HYPERTENSIONAHA.109.145409. Epub 2009 Dec 7. PMID 19996061
- [Background] Liu Z, Liu J, Jahn LA, Fowler DE, Barrett EJ. Infusing lipid raises plasma free fatty acids and induces insulin resistance in muscle microvasculature. J Clin Endocrinol Metab. 2009 Sep;94(9):3543-9. doi: 10.1210/jc.2009-0027. Epub 2009 Jun 30. PMID 19567533
- [Background] Liu J, Jahn LA, Fowler DE, Barrett EJ, Cao W, Liu Z. Free fatty acids induce insulin resistance in both cardiac and skeletal muscle microvasculature in humans. J Clin Endocrinol Metab. 2011 Feb;96(2):438-46. doi: 10.1210/jc.2010-1174. Epub 2010 Nov 3. PMID 21047922
- [Background] Vincent MA, Barrett EJ, Lindner JR, Clark MG, Rattigan S. Inhibiting NOS blocks microvascular recruitment and blunts muscle glucose uptake in response to insulin. Am J Physiol Endocrinol Metab. 2003 Jul;285(1):E123-9. doi: 10.1152/ajpendo.00021.2003. PMID 12791603
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Youd JM, Rattigan S, Clark MG. Acute impairment of insulin-mediated capillary recruitment and glucose uptake in rat skeletal muscle in vivo by TNF-alpha. Diabetes. 2000 Nov;49(11):1904-9. doi: 10.2337/diabetes.49.11.1904. PMID 11078458
- [Background] Liu Z. The vascular endothelium in diabetes and its potential as a therapeutic target. Rev Endocr Metab Disord. 2013 Mar;14(1):1-3. doi: 10.1007/s11154-013-9238-8. No abstract available. PMID 23397463
- [Background] Gavin TP, Stallings HW 3rd, Zwetsloot KA, Westerkamp LM, Ryan NA, Moore RA, Pofahl WE, Hickner RC. Lower capillary density but no difference in VEGF expression in obese vs. lean young skeletal muscle in humans. J Appl Physiol (1985). 2005 Jan;98(1):315-21. doi: 10.1152/japplphysiol.00353.2004. Epub 2004 Aug 6. PMID 15298982
- [Background] Lillioja S, Young AA, Culter CL, Ivy JL, Abbott WG, Zawadzki JK, Yki-Jarvinen H, Christin L, Secomb TW, Bogardus C. Skeletal muscle capillary density and fiber type are possible determinants of in vivo insulin resistance in man. J Clin Invest. 1987 Aug;80(2):415-24. doi: 10.1172/JCI113088. PMID 3301899
- [Background] Solomon TP, Haus JM, Li Y, Kirwan JP. Progressive hyperglycemia across the glucose tolerance continuum in older obese adults is related to skeletal muscle capillarization and nitric oxide bioavailability. J Clin Endocrinol Metab. 2011 May;96(5):1377-84. doi: 10.1210/jc.2010-2069. Epub 2011 Feb 2. PMID 21289242
- [Background] Olsson AK, Dimberg A, Kreuger J, Claesson-Welsh L. VEGF receptor signalling - in control of vascular function. Nat Rev Mol Cell Biol. 2006 May;7(5):359-71. doi: 10.1038/nrm1911. PMID 16633338
- [Background] Tang K, Breen EC, Gerber HP, Ferrara NM, Wagner PD. Capillary regression in vascular endothelial growth factor-deficient skeletal muscle. Physiol Genomics. 2004 Jun 17;18(1):63-9. doi: 10.1152/physiolgenomics.00023.2004. Epub 2004 Jun 17. PMID 15084712
- [Background] Bonner JS, Lantier L, Hasenour CM, James FD, Bracy DP, Wasserman DH. Muscle-specific vascular endothelial growth factor deletion induces muscle capillary rarefaction creating muscle insulin resistance. Diabetes. 2013 Feb;62(2):572-80. doi: 10.2337/db12-0354. Epub 2012 Sep 21. PMID 23002035
- [Background] Hazarika S, Dokun AO, Li Y, Popel AS, Kontos CD, Annex BH. Impaired angiogenesis after hindlimb ischemia in type 2 diabetes mellitus: differential regulation of vascular endothelial growth factor receptor 1 and soluble vascular endothelial growth factor receptor 1. Circ Res. 2007 Oct 26;101(9):948-56. doi: 10.1161/CIRCRESAHA.107.160630. Epub 2007 Sep 6. PMID 17823371
- [Background] Roque FR, Hernanz R, Salaices M, Briones AM. Exercise training and cardiometabolic diseases: focus on the vascular system. Curr Hypertens Rep. 2013 Jun;15(3):204-14. doi: 10.1007/s11906-013-0336-5. PMID 23519745
- [Background] Castorena CM, Arias EB, Sharma N, Cartee GD. Postexercise improvement in insulin-stimulated glucose uptake occurs concomitant with greater AS160 phosphorylation in muscle from normal and insulin-resistant rats. Diabetes. 2014 Jul;63(7):2297-308. doi: 10.2337/db13-1686. Epub 2014 Mar 7. PMID 24608437
- [Background] Vincent MA, Clerk LH, Lindner JR, Price WJ, Jahn LA, Leong-Poi H, Barrett EJ. Mixed meal and light exercise each recruit muscle capillaries in healthy humans. Am J Physiol Endocrinol Metab. 2006 Jun;290(6):E1191-7. doi: 10.1152/ajpendo.00497.2005. PMID 16682488
- [Background] Inyard AC, Clerk LH, Vincent MA, Barrett EJ. Contraction stimulates nitric oxide independent microvascular recruitment and increases muscle insulin uptake. Diabetes. 2007 Sep;56(9):2194-200. doi: 10.2337/db07-0020. Epub 2007 Jun 11. PMID 17563063
- [Background] Richter EA, Hargreaves M. Exercise, GLUT4, and skeletal muscle glucose uptake. Physiol Rev. 2013 Jul;93(3):993-1017. doi: 10.1152/physrev.00038.2012. PMID 23899560
- [Background] Wheatley CM, Rattigan S, Richards SM, Barrett EJ, Clark MG. Skeletal muscle contraction stimulates capillary recruitment and glucose uptake in insulin-resistant obese Zucker rats. Am J Physiol Endocrinol Metab. 2004 Oct;287(4):E804-9. doi: 10.1152/ajpendo.00077.2004. Epub 2004 Jun 22. PMID 15213062
- [Background] Hoier B, Hellsten Y. Exercise-induced capillary growth in human skeletal muscle and the dynamics of VEGF. Microcirculation. 2014 May;21(4):301-14. doi: 10.1111/micc.12117. PMID 24450403
- [Background] Olfert IM, Howlett RA, Tang K, Dalton ND, Gu Y, Peterson KL, Wagner PD, Breen EC. Muscle-specific VEGF deficiency greatly reduces exercise endurance in mice. J Physiol. 2009 Apr 15;587(Pt 8):1755-67. doi: 10.1113/jphysiol.2008.164384. Epub 2009 Feb 23. PMID 19237429
- [Background] Basu A, Charkoudian N, Schrage W, Rizza RA, Basu R, Joyner MJ. Beneficial effects of GLP-1 on endothelial function in humans: dampening by glyburide but not by glimepiride. Am J Physiol Endocrinol Metab. 2007 Nov;293(5):E1289-95. doi: 10.1152/ajpendo.00373.2007. Epub 2007 Aug 21. PMID 17711996
- [Background] Aronis KN, Chamberland JP, Mantzoros CS. GLP-1 promotes angiogenesis in human endothelial cells in a dose-dependent manner, through the Akt, Src and PKC pathways. Metabolism. 2013 Sep;62(9):1279-86. doi: 10.1016/j.metabol.2013.04.010. Epub 2013 May 14. PMID 23684008
- [Background] Jayaweera AR, Wei K, Coggins M, Bin JP, Goodman C, Kaul S. Role of capillaries in determining CBF reserve: new insights using myocardial contrast echocardiography. Am J Physiol. 1999 Dec;277(6):H2363-72. doi: 10.1152/ajpheart.1999.277.6.H2363. PMID 10600857
- [Background] Laine H, Nuutila P, Luotolahti M, Meyer C, Elomaa T, Koskinen P, Ronnemaa T, Knuuti J. Insulin-induced increment of coronary flow reserve is not abolished by dexamethasone in healthy young men. J Clin Endocrinol Metab. 2000 May;85(5):1868-73. doi: 10.1210/jcem.85.5.6597. PMID 10843167
- [Background] Laine H, Sundell J, Nuutila P, Raitakari OT, Luotolahti M, Ronnemaa T, Elomaa T, Koskinen P, Knuuti J. Insulin induced increase in coronary flow reserve is abolished by dexamethasone in young men with uncomplicated type 1 diabetes. Heart. 2004 Mar;90(3):270-6. doi: 10.1136/hrt.2003.013722. PMID 14966043
- [Background] Sundell J, Nuutila P, Laine H, Luotolahti M, Kalliokoski K, Raitakari O, Knuuti J. Dose-dependent vasodilating effects of insulin on adenosine-stimulated myocardial blood flow. Diabetes. 2002 Apr;51(4):1125-30. doi: 10.2337/diabetes.51.4.1125. PMID 11916935
- [Background] Sundell J, Laine H, Nuutila P, Ronnemaa T, Luotolahti M, Raitakari O, Knuuti J. The effects of insulin and short-term hyperglycaemia on myocardial blood flow in young men with uncomplicated Type I diabetes. Diabetologia. 2002 Jun;45(6):775-82. doi: 10.1007/s00125-002-0819-4. Epub 2002 Apr 25. PMID 12107720
- [Background] Chai W, Liu J, Jahn LA, Fowler DE, Barrett EJ, Liu Z. Salsalate attenuates free fatty acid-induced microvascular and metabolic insulin resistance in humans. Diabetes Care. 2011 Jul;34(7):1634-8. doi: 10.2337/dc10-2345. Epub 2011 May 26. PMID 21617098
- [Background] Zhao T, Parikh P, Bhashyam S, Bolukoglu H, Poornima I, Shen YT, Shannon RP. Direct effects of glucagon-like peptide-1 on myocardial contractility and glucose uptake in normal and postischemic isolated rat hearts. J Pharmacol Exp Ther. 2006 Jun;317(3):1106-13. doi: 10.1124/jpet.106.100982. Epub 2006 Feb 17. PMID 16489128
- [Background] Bose AK, Mocanu MM, Carr RD, Brand CL, Yellon DM. Glucagon-like peptide 1 can directly protect the heart against ischemia/reperfusion injury. Diabetes. 2005 Jan;54(1):146-51. doi: 10.2337/diabetes.54.1.146. PMID 15616022
- [Background] Nikolaidis LA, Mankad S, Sokos GG, Miske G, Shah A, Elahi D, Shannon RP. Effects of glucagon-like peptide-1 in patients with acute myocardial infarction and left ventricular dysfunction after successful reperfusion. Circulation. 2004 Mar 2;109(8):962-5. doi: 10.1161/01.CIR.0000120505.91348.58. Epub 2004 Feb 23. PMID 14981009